CLINICAL TRIAL: NCT00305188
Title: A Multicenter, Randomized Double-blind Placebo Controlled Phase III Study of the Efficacy of Xaliproden in Preventing the Neurotoxicity of Oxaliplatin in First-line Treatment of Patients With Metastatic Colorectal Cancer Treated With Oxaliplatin / 5-FU/LV
Brief Title: Evaluation of the Efficacy of Xaliproden (SR57746A) in Preventing the Neurotoxicity of Oxaliplatin / 5FU/LV Chemotherapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EFC5505; EUDRACT : 2005-002570-30
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-04

CONDITIONS: Metastases; Colorectal Neoplasms; Colorectal Carcinoma
Keywords: Neurotoxicity syndromes; Paresthesia; Oxaliplatin; Xaliproden
MeSH Terms: conditions — Neoplasm Metastasis; Colorectal Neoplasms; Neurotoxicity Syndromes; Paresthesia | interventions — xaliproden; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Xaliproden (SR57746A) (Experimental)
  Interventions: Drug: Xaliproden (SR57746A); Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Oxaliplatin; Drug: 5-Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Xaliproden (SR57746A) — oral administration
  Arms: Xaliproden (SR57746A)
Drug: Placebo — oral administration
  Arms: Placebo
Drug: Oxaliplatin — IV administration
Drug: 5-Fluorouracil — IV administration
  Other Names: 5-FU
Drug: Leucovorin — IV administration
  Other Names: LV

SUMMARY:
Primary Objective : Compare the risk of occurrence of Grade3-4 cumulative peripheral sensory neuropathy (PSN) relative to cumulative dose of oxaliplatin between treatment group and placebo group.

Main Secondary Objective : Compare the response rate (RR) between treatment group and placebo group in order to ensure that the efficacy of the chemotherapy is not compromised by the addition of xaliproden to the chemotherapeutic regimen.

Other Secondary Objectives : study of the neurotoxicity parameters (Duration of oxaliplatin-induced PSN (G2,3,4); overall incidence of PSN during treatment; dose of onset of PSN ; incidence of dose-reduction and dose delay due to PSN; incidence of oxaliplatin treatment discontinuation due to PSN; change in Nerve Conduction Studies (NCS)) ; study of the safety profile (other than PSN) ; study of the chemotherapy efficacy (progression free survival, overall survival).

ELIGIBILITY:
Inclusion Criteria:

Main inclusion criteria :

* Histologically or cytologically-proven metastatic cancer of the colon or rectum.
* Metastatic disease not amenable to potentially curative treatment (eg: inoperable metastatic disease).
* Male or female aged >18 years.
* WHO Performance Status (PS) : 0 or 1.
* Measurable disease.
* No prior chemotherapeutic regimen for metastatic disease.
* Disease-free interval from end of adjuvant therapy of at least 6 months (1 year if oxaliplatin was part of the adjuvant therapy).
* Prior radiotherapy is permitted if it was not administered to target lesions identified for this study - unless progression within the radiation portal is documented - and provided it has been completed at least 3 weeks before randomization.
* Signed written informed consent prior to study entry.

Exclusion Criteria:

Main exclusion criteria :

* Any condition or past medical history that contra-indicates treatment with oxaliplatin and 5-FU, as reported in approved labeling information.
* Received chemotherapeutic agents other than 5-FU, LV, Levamisole, irinotecan, capecitabine, oxaliplatin as part of adjuvant therapy.
* Peripheral neuropathy >Grade 1.
* Concomitant treatments with drugs/ingredients reported to have a potential activity in preventing peripheral sensory neuropathy.
* Concurrent active cancer originating from a primary site other than colon or rectum.
* Presence of any symptom suggesting brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of peripheral sensory neuropathy using the Oxaliplatin specific scale for dose adjustment | Q2W during treatment, Q4W to Q12W during post-treatment follow-up

SECONDARY OUTCOMES:
Main: response rate using RECIST criteria | Q8W
Other: nerve conduction studies | baseline, end of treatment with oxaliplatin, end of treatment with study drug
Other: progression free survival and survival | Q8W and study period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (13):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Liu J, Wang X, Sahin IH, Imanirad I, Felder SI, Kim RD, Xie H. Tumor Response-speed Heterogeneity as a Novel Prognostic Factor in Patients With Metastatic Colorectal Cancer. Am J Clin Oncol. 2023 Feb 1;46(2):50-57. doi: 10.1097/COC.0000000000000972. Epub 2022 Dec 26. PMID 36606664
- [Derived] Abdel-Rahman O. Effect of Body Mass Index on 5-FU-Based Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer; A Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Dec;18(4):e385-e393. doi: 10.1016/j.clcc.2019.07.005. Epub 2019 Jul 15. PMID 31378656
- [Derived] Abdel-Rahman O. Impact of Sex on Chemotherapy Toxicity and Efficacy Among Patients With Metastatic Colorectal Cancer: Pooled Analysis of 5 Randomized Trials. Clin Colorectal Cancer. 2019 Jun;18(2):110-115.e2. doi: 10.1016/j.clcc.2018.12.006. Epub 2018 Dec 28. PMID 30679026